CLINICAL TRIAL: NCT06970457
Title: The Interaction of Body Composition, Sex Hormones and Exercise in Men
Acronym: AHA-NWO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oklahoma State University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-24-542
Record Dates: First submitted 2025-03-14; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Normal-weight Obesity
Keywords: body composition; sex hormones; exercise; metabolic health
MeSH Terms: conditions — Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Resistance Exercise Training (Experimental): 12-weeks of progressive and individualized resistance exercise training
  Interventions: Behavioral: Resistance Exercise Training; Behavioral: Aerobic Exercise Training
- Aerobic Exercise Training (Active Comparator): 12-weeks of progressive and individualized aerobic exercise training
  Interventions: Behavioral: Resistance Exercise Training; Behavioral: Aerobic Exercise Training

INTERVENTIONS:
Behavioral: Resistance Exercise Training — 12-week progressive and individualized resistance exercise training program
Behavioral: Aerobic Exercise Training — 12-week progressive and individualized aerobic exercise training program

SUMMARY:
The overall objective of this project is to advance understanding of the causes of normal weight obesity (NWO) in men, namely the hormone profile and related potential mediating mechanisms, and the efficacy of different modes of exercise to restore body composition and cardiometabolic health in this population.

ELIGIBILITY:
Inclusion Criteria:

* Biological male
* BMI 18.5 - 24.9 kg/m2 or >/= 30 kg/m2
* Body fat <20% or >/= 25%
* Ability and willingness to engage in an exercise training regimen

Exclusion Criteria:

* Presence of a chronic health condition, or regular use of associate prescribed medications, that would substantially impact study variables
* Excessive alcohol use or use of tobacco products, vape products, or illicit drugs
* Presence of an electrical implant, such as a pacemaker

Ages: 18 Years to 79 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Fat Mass | Baseline/enrollment only in control participants; Baseline/enrollment/pre-intervention and post-intervention (12 weeks after baseline testing) in intervention participants
  Fat mass, measured in kg and as a percentage of total body mass Measured through dual-energy X ray absorptiometry
Lean mass | Baseline/enrollment only in control participants; Baseline/enrollment/pre-intervention and post-intervention (12 weeks after baseline testing) in intervention participants
  Lean mass, measured in kg and as a percentage of total body mass Measured through dual-energy X ray absorptiometry
Testosterone | Baseline/enrollment only in control participants; Baseline/enrollment/pre-intervention and post-intervention (12 weeks after baseline testing) in intervention participants
  Human testosterone, measured in serum via Novus Biologicals Human Testosterone ELISA Kit (Colorimetric). Measured in pg/mL.
Human Growth Hormone | Baseline/enrollment only in control participants; Baseline/enrollment/pre-intervention and post-intervention (12 weeks after baseline testing) in intervention participants
  Human Growth Hormone (HGH), measured in serum via R&D Systems™ Human Growth Hormone Quantikine ELISA Kit Measured in pg/mL
Estradiol | Baseline/enrollment only in control participants; Baseline/enrollment/pre-intervention and post-intervention (12 weeks after baseline testing) in intervention participants
  Human estradiol, measured in serum via Novus Biologicals Human Estradiol ELISA Kit (Colorimetric); measured in pg/mL
SHBG | Baseline/enrollment only in control participants; Baseline/enrollment/pre-intervention and post-intervention (12 weeks after baseline testing) in intervention participants
  Sex Hormone Binding Globulin (SHBG), measured in serum via R&D Systems™ Human SHBG Quantikine ELISA Kit; measured in pg/mL
Luteinizing Hormone | Baseline/enrollment only in control participants; Baseline/enrollment/pre-intervention and post-intervention (12 weeks after baseline testing) in intervention participants
  Luteinizing Hormone (LH), measured in serum via Invitrogen™ Luteinizing Hormone Human ELISA Kit; measured in pg/mL
FSH | Baseline/enrollment only in control participants; Baseline/enrollment/pre-intervention and post-intervention (12 weeks after baseline testing) in intervention participants
  Follicle Stimulating Hormone (FSH), measured in serum via Invitrogen™ Human FSH ELISA Kit; measured in pg/mL
Adiponectin | Baseline/enrollment only in control participants; Baseline/enrollment/pre-intervention and post-intervention (12 weeks after baseline testing) in intervention participants
  Adiponectin, measured in serum via Invitrogen™ Adiponectin Human ELISA Kit; measured in pg/mL
Leptin | Baseline/enrollment only in control participants; Baseline/enrollment/pre-intervention and post-intervention (12 weeks after baseline testing) in intervention participants
  Leptin, measured in serum via Invitrogen™ Leptin Human ELISA Kit; measured in pg/mL
Aromatase | Baseline/enrollment only in control participants; Baseline/enrollment/pre-intervention and post-intervention (12 weeks after baseline testing) in intervention participants
  Aromatase enzyme, measured in serum via Invitrogen™ Human Aromatase ELISA Kit; measured in ng/mL
Insulin | Baseline/enrollment only in control participants; Baseline/enrollment/pre-intervention and post-intervention (12 weeks after baseline testing) in intervention participants
  Insulin, measured in serum via Eagle Biosciences Inc Insulin Ultrasensitive ELISA; measured in mU/L
KISS1 | Baseline/enrollment only in control participants; Baseline/enrollment/pre-intervention and post-intervention (12 weeks after baseline testing) in intervention participants
  Kisspeptin (KISS1), measured in serum via Biomatik Corporation Human Kisspeptin 1 (KISS1) ELISA Kit; measured in pg/mL
GnRH | Baseline/enrollment only in control participants; Baseline/enrollment/pre-intervention and post-intervention (12 weeks after baseline testing) in intervention participants
  Gonadotropin-releasing hormone (GnRH), measured in serum via Biomatik Corporation Human Gonadotropin Releasing Hormone (GnRH) ELISA Kit; measured in pg/mL
Inflammatory Cytokine Panel | Baseline/enrollment only in control participants; Baseline/enrollment/pre-intervention and post-intervention (12 weeks after baseline testing) in intervention participants
  Human High Sensitivity T-Cell 15-Plex Discovery Assay®, conducted by Eve Technologies, that includes GM-CSF, IFN-γ, IL-1β, IL-1RA, IL-2, IL-4, IL-5, IL-6, IL-8, IL-10, IL-12p40, IL-12p70, IL-13, MCP-1 and TNFα; measured in pg/mL
Triglycerides | Baseline/enrollment only in control participants; Baseline/enrollment/pre-intervention and post-intervention (12 weeks after baseline testing) in intervention participants
  Triglycerides, measured in whole blood via Piccolo Xpress clinical chemistry analyzer with Lipid Panel Plus reagent discs; measured in mg/dL
Glucose | Baseline/enrollment only in control participants; Baseline/enrollment/pre-intervention and post-intervention (12 weeks after baseline testing) in intervention participants
  Glucose, measured in whole blood via Piccolo Xpress clinical chemistry analyzer with Lipid Panel Plus reagent discs; measured in mg/dL
HDL-C | Baseline/enrollment only in control participants; Baseline/enrollment/pre-intervention and post-intervention (12 weeks after baseline testing) in intervention participants
  High-density Lipoprotein Cholesterol (HDL-C), measured in whole blood via Piccolo Xpress clinical chemistry analyzer with Lipid Panel Plus reagent discs; measured in mg/dL
Total Cholesterol | Baseline/enrollment only in control participants; Baseline/enrollment/pre-intervention and post-intervention (12 weeks after baseline testing) in intervention participants
  Total Cholesterol, measured in whole blood via Piccolo Xpress clinical chemistry analyzer with Lipid Panel Plus reagent discs; measured in mg/dL
Visceral Adipose Tissue | Baseline/enrollment only in control participants; Baseline/enrollment/pre-intervention and post-intervention (12 weeks after baseline testing) in intervention participants
  Visceral Adipose Tissue (VAT), measured in g and g/cm3 via dual-energy X ray absorptiometry

SECONDARY OUTCOMES:
ALT | Baseline/enrollment only in control participants; Baseline/enrollment/pre-intervention and post-intervention (12 weeks after baseline testing) in intervention participants
  Alanine Transaminase (ALT) liver enzyme, measured in whole blood via Piccolo Xpress clinical chemistry analyzer with Lipid Panel Plus reagent discs; measured in U/L
AST | Baseline/enrollment only in control participants; Baseline/enrollment/pre-intervention and post-intervention (12 weeks after baseline testing) in intervention participants
  Aspartate Aminotransferase (AST), measured in whole blood via Piccolo Xpress clinical chemistry analyzer with Lipid Panel Plus reagent discs; measured in U/L
Bone Mineral Density | Baseline/enrollment only in control participants; Baseline/enrollment/pre-intervention and post-intervention (12 weeks after baseline testing) in intervention participants
  Whole-body Bone Mineral Density (BMD), measured via dual-energy X ray absorptiometry; measured in g/cm3
Height | Baseline/enrollment
  Height, measured in inches via portable stadiometer
Body Mass | Baseline/enrollment only in control participants; Baseline/enrollment/pre-intervention and post-intervention (12 weeks after baseline testing) in intervention participants
  Body mass, measured in kg via Seca mBCA (medical body composition analyzer) 514
Waist Circumference | Baseline/enrollment only in control participants; Baseline/enrollment/pre-intervention and post-intervention (12 weeks after baseline testing) in intervention participants
  Waist Circumference, measured in inches via standard Gulick tape measure.
Free-living Dietary Intake | Baseline/enrollment only in control participants; Baseline/enrollment/pre-intervention and post-intervention (12 weeks after baseline testing) in intervention participants
  Free-Living Dietary Intake, measured via 3-day food record. Participant completes the record for 3 days and returns to the researchers.
Free-living Physical Activity | Baseline/enrollment only in control participants; Baseline/enrollment/pre-intervention and post-intervention (12 weeks after baseline testing) in intervention participants
  Free-living Physical Activity, assessed through accelerometry via Actigraph wGT3X-BT accelerometers. Participant wears the accelerometer for 3 days, then returns it to the researchers.
Aerobic Capacity | Baseline/enrollment only in control participants; Baseline/enrollment/pre-intervention and post-intervention (12 weeks after baseline testing) in intervention participants
  Aerobic Capacity, also known as VO2peak, assessed via YMCA submaximal exercise test, completed on a cycle ergometer.
Resting Energy Expenditure | Baseline/enrollment only in control participants; Baseline/enrollment/pre-intervention and post-intervention (12 weeks after baseline testing) in intervention participants
  Resting Energy Expenditure (REE), measured via indirect calorimetry. The test is conducted with a Parvo Medics True One 2400 metabolic analysis system with a canopy hood; measured as kcal/day.
Upper-body Muscle Strength | Baseline/enrollment only in control participants; Baseline/enrollment/pre-intervention and post-intervention (12 weeks after baseline testing) in intervention participants
  Upper-body Muscle Strength, measured via three-repetition maximum (3RM) bench press; measured in pounds.
Lower-body Muscle Strength | Baseline/enrollment only in control participants; Baseline/enrollment/pre-intervention and post-intervention (12 weeks after baseline testing) in intervention participants
  Lower-body Muscle Strength, measured via knee extensor test with a Biodex dynamometer and three-repetition maximum (3RM) leg press exercise; measured as peak torque in Nm and pounds, respectively.
Upper-body Muscle Power | Baseline/enrollment only in control participants; Baseline/enrollment/pre-intervention and post-intervention (12 weeks after baseline testing) in intervention participants
  Upper-body Muscle Power, measured via seated medicine ball toss; measured in inches (thrown).
Lower-body Muscle Power | Baseline/enrollment only in control participants; Baseline/enrollment/pre-intervention and post-intervention (12 weeks after baseline testing) in intervention participants
  Lower-body Muscle Power, measured via maximal voluntary contraction of the knee extensors with a Biodex dynamometer; measured as peak torque in Nm.
Blood Pressure | Baseline/enrollment only in control participants; Baseline/enrollment/pre-intervention and post-intervention (12 weeks after baseline testing) in intervention participants
  Blood Pressure, both systolic and diastolic, measured with an automated blood pressure cuff; measured in mmHg.

CONTACTS AND LOCATIONS:
Overall Officials: Sam Emerson, PhD, Principal Investigator — Oklahoma State University
Locations (1):
- Oklahoma State University, Stillwater, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Undecided